CLINICAL TRIAL: NCT03397784
Title: Can Respiratory Variation in Inferior Vena Cava Diameter After Tidal Volume Challenge Predict Fluid Responsiveness in Cardiac Surgical Patients With Mechanical Ventilation
Brief Title: IVC Variation After VT Challenge to Predict Fluid Responsiveness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: VIVC-TVC
Record Dates: First submitted 2018-01-01; First posted 2018-01-12 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Cardiac Surgery; Fluid Challenge; Fluid Responsiveness; Mechanical Ventilation
Keywords: Tidal volume challenge; Fluid responsiveness; Preload responsiveness; Functional hemodynamic monitoring; Cardiac surgery; inferior vena cava variation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- fluid responders: Patients whose stroke volume index increase by ≥15% in response to a 500-ml fluid bolus was defined as fluid responders.
- fluid non-responders: Patients whose stroke volume index increase by <15% in response to a 500-ml fluid bolus was defined as fluid non-responders.

SUMMARY:
The purpose of the study was to evaluate the efficacy of using the respiratory variation in inferior vena cava diameters as an index of fluid responsiveness after tidal volume challenge in mechanically ventilated patients after cardiac surgery.

DETAILED DESCRIPTION:
The "tidal volume challenge" is a novel test to predict fluid responsiveness in patents in shock, ventilated using low tidal volume without spontaneous breathing activity. The test involves transiently increasing tidal volume from 8 ml/kg PBW to 12 ml/kg PBW for one minute and observing the change in PPV or SVV. The aim of this study was to evaluate whether the respiratory variation in inferior vena cava diameter after tidal volume challenge can predict fluid responsiveness in cardiac surgical patients with mechanical ventilation

ELIGIBILITY:
Inclusion Criteria:

* acute circulatory failure (low blood pressure or urine output, tachycardia, or mottling)
* clinical signs of organ hypoperfusion (renal dysfunction or hyperlactatemia)

Exclusion Criteria:

* a contraindication to elevation of tidal volume
* evidence of cardiac arrhythmia
* left ventricular ejection fraction less than 50%
* echocardiographic examination that showed the existence of severe tricuspid or mitral regurgitation or right heart dysfunction
* intracardiac shunt
* pulmonary hypertension
* severe chronic obstructive pulmonary disease
* a contraindication to the passive leg raising (PLR) test
* air leakage through chest drains
* abdominal compartment syndrome
* portal hypertension
* pregnancy
* inability to perform ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after cardiac surgery
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-02-03 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
fluid responsiveness | after fluid challenge (30min)
  Patients will be classified as "fluid responders" if there is an increase in SV ≥15% after the fluid challenge, and the remaining patients are classified as "fluid non-responders"

SECONDARY OUTCOMES:
inferior vena cava variation | After tidal volume challenge (1 minute) and fluid challenge (30 minute)
  Ultrasound equipment with convex probe will be used to measure IVC diameters of the patients in supine position.The IVC sagittal section is described with the probe in the area of subxiphoid. IVC diameters at the junction point of the IVC and right atrium (2cm caudal) are standardized measurement. The maximum anterior-posterior dimension came out from end-inspiration (IVCi, mm), whereas the minimum IVC diameter was shown in end-expiration (IVCe, mm). The IVC variation (IVCV) is calculated using the formula: IVCV (%) = (IVCi - IVCe) / [(IVCi+ IVCe) / 2] ×100%.

CONTACTS AND LOCATIONS:
Overall Officials: Tu Guo-wei, PhD, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China